CLINICAL TRIAL: NCT04406142
Title: Surfactant Administration Via Thin Catheter Using a Specially Adapted Video Laryngoscope - a Prospective, Multicenter Trial, Assessing the Feasibility of the VISUAL Method (Video Surfactant Administration Laryngoscopy)
Brief Title: Surfactant Administration Via Thin Catheter Using a Specially Adapted Video Laryngoscope - the VISUAL Method
Acronym: VISUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Dany Waisman, Director of the Newborn Unit Department of Neonatology, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMC-17-0007-CTIL
Record Dates: First submitted 2020-02-10; First posted 2020-05-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: respiratory distress syndrome; videolaryngoscopy; newborn infant; premature newborn infant; surfactant administration
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment feasibility (Experimental): feasibility, safety and effectiveness assessment
  Interventions: Device: VISUAL

INTERVENTIONS:
Device: VISUAL — thin catheter insertion between vocal cords under direct specially adapted videolaryngoscopy

SUMMARY:
Surfactant administration via thin catheter using a specially adapted video laryngoscope - a prospective, multicenter trial, assessing the feasibility of the VISUAL method (Video Surfactant Administration Laryngoscopy).

The study will search for the number of attempts until surfactant is administrated, assessment of the infants' stability during the procedure, duration of the entire procedure, form laryngoscope insertion to surfactant administration.

DETAILED DESCRIPTION:
In this study the investigators intend to assess the feasibility of surfactant administration via a thin catheter using a specially adapted video laryngoscope, with a groove designed to allow insertion of an endovascular catheter without the use of other instruments in the oral cavity (forceps ect.).

The laryngoscope is manufactured by Peak Medic Ltd, Natania, Israel.

Primary Endpoints

1. - Number of attempts until surfactant is administrated
2. - Assessment of the infants' stability during the procedure - saturation, bradycardia, tachycardia.
3. - Duration of the entire procedure, form laryngoscope insertion to surfactants administration.

4. Secondary Endpoints

1. - Need of invasive mechanical ventilation in the next 24 hours.
2. - Complications reports
3. - Subjective procedure scale of assessment
4. - Unexpected pitfalls reports
5. - Safety assessment of the procedure

ELIGIBILITY:
Inclusion Criteria:

1. - Premature infants with gestational age 30-36 weeks.
2. - Diagnosis of respiratory distress syndrome
3. - Spontaneously breathing with non-invasive positive pressure ventilation.
4. - Maximal age 3 days.

Exclusion Criteria:

1. - Apgar score at 5 min < 5
2. - Need for chest compressions or medication upon delivery.
3. - Evident major congenital malformation, metabolic or genetic disorders.
4. - Clinical evidence of sepsis.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures | 1 year
  Success for surfactant administration - yes / no

SECONDARY OUTCOMES:
Secondary outcome measures 1 | 1 year
  Assessment of the infants' SPO2 %
Secondary outcome measures 2 | 1 year
  Heart rate during the procedure
Secondary outcome measures 3 | 1 year
  Respiratory rate (breaths per minute)
Secondary outcome measures 4 | 1 year
  number of attempts for vocal cords visualization (number)
Secondary outcome measures 5 | 1 year
  Duration of the procedure (seconds)
Secondary outcome measures 6 | 1 year
  Need for mechanical ventilaton witin 24 hours following procedure (yes-no)

CONTACTS AND LOCATIONS:
Overall Officials: Dan I Waisman, MD, Principal Investigator — Department of Neonatology, Carmel Medical Center
Locations (1):
- Department of Neonatology, Carmel Medical Center, Haifa, Israel